CLINICAL TRIAL: NCT06501898
Title: Tributyrin: Time Course & Efficacy to Improve Health & Performance
Acronym: CoreBiome
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Loss of funding
Sponsor: Florida State University (Other)
Collaborators: Compound Solutions Inc. (Industry)
Responsible Party: Principal Investigator, Michael J. Ormsbee, Professor, Florida State University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: STUDY00004764
Record Dates: First submitted 2024-06-27; First posted 2024-07-15 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Metabolite Concentration; Gut Permeability; Inflammation; Sleep; Performance
MeSH Terms: conditions — Inflammation | interventions — tributyrin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CoreBiome (Active Comparator): Participants will be given tributyrin (as CoreBiome)
  Interventions: Dietary Supplement: CoreBiome
- Placebo (Placebo Comparator): Participants will be given a taste-, color-, and odor-matched placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: CoreBiome — 300 mg, once daily of tributyrin for 4 weeks
  Other Names: Tributyrin
  Arms: CoreBiome
Dietary Supplement: Placebo — 300 mg, once daily of placebo for 4 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if tributyrin supplementation improves metabolite concentrations, overall health biomarkers, and performance in sedentary men and women. The study would further understand the potential usage of tributyrin as a health and performance increasing supplement through improving gut and immune health, sleep, and performance as well as reduce inflammation. Participants will supplement for tributyrin for 4 weeks and complete fecal metabolite measures, cardiovascular evaluation, sleep assessment, and exercise testing as well as provide blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Age: 30-50 years
* Sedentary (<150 minutes of aerobic exercise per week)

Exclusion Criteria:

* Chronic, uncontrolled metabolic, cardiovascular, gastrointestinal, or hepatic disease
* Consumption of supplements known to impact the microbiome, hydration status, core temperature, or exercise performance
* Experienced previous heat illness
* Known injuries that limit exercise
* BMI ≥ 40 kg/m^2
* Pregnant

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2024-08-19 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Metabolite Concentration | 2 and 4 weeks after onset of CoreBiome supplementation; 2 and 4 weeks after onset of Placebo supplementation
  Fecal butyrate concentration

SECONDARY OUTCOMES:
Gut permeability | 10 minutes before and 5 minutes prior to completion of exercise bout (i.e., mid-exercise)
  Urine dual sugar absorption, Plasma sCD14
Inflammation | 10 minutes before and 5 minutes prior to completion of exercise bout (i.e., mid-exercise)
  Whole-body inflammation (IL-6 and IL-10) and gut-specific inflammation (IL-17 and IL-23)
Immune cell composition | 10 minutes before and 5 minutes prior to completion of exercise bout (i.e., mid-exercise)
  Relative proportions of serum immune cells (e.g., macrophages, neutrophils, T cells, B cells, etc.)
Sleep Quality | Four weeks prior to day of exercise bout
  Number of sleep disturbances
Sleep quantity | Four weeks prior to day of exercise bout
  Sleep duration
Substrate Utilization (mid-exercise) | During exercise bout
  Respiratory exchange ratio assessment via metabolic testing during cycling exercise
Perceived exertion (mid-exercise) | During exercise bout
  Subjective perceived exertion survey during cycling exercise
Total completed distance (mid-exercise) | During exercise bout
  Total completed distance during cycling exercise
Maximum sprint power (mid-exercise) | During exercise bout
  Maximum power quantification during cycling exercise
Average sprint power (mid-exercise) | During exercise bout
  Average power quantification during cycling exercise

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Sports Sciences & Medicine, Tallahassee, Florida, United States